CLINICAL TRIAL: NCT04992715
Title: A Single-arm, Phase II Study to Evaluate PD-L1 Expression in Non-Small Cell Lung Cancer Using the 99mTc Labelled Anti-PD-L1 Single Domain Antibody (NM-01)
Brief Title: PD-L1 Expression in Lung Cancer
Acronym: PELICAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NanoMab Technology (UK) Limited (Industry)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PELICAN; 2020-002809-26 (EudraCT Number)
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: PD-L1 Expression; Immunohistochemistry; SPECT/CT Imaging; Molecular Imaging; Heterogeneity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic Non-Small Cell Lung Cancer (Experimental): Subjects with metastatic non-small cell lung cancer will be recruited as per protocol inclusion/exclusion criteria and will undergo [99mTc]-anti-PDL1 single-domain antibody ([99mTc]-NM-01) SPECT/CT imaging.
  [99mTc]-NM-01 SPECT/CT images will be compared to immunohistochemistry PD-L1 expression results.
  Interventions: Diagnostic Test: [99mTc]-NM01 SPECT/CT

INTERVENTIONS:
Diagnostic Test: [99mTc]-NM01 SPECT/CT — Technetium-99m radiolabelled anti-PD-L1 single-domain antibody (NM01) single-photon emission computed tomography (SPECT)/computed tomography (CT)

SUMMARY:
This study will measure PD-L1 expression in metastatic NSCLC (primary tumour and metastatic lesions) using [99mTc]-NM-01 SPECT/CT and compare to PD-L1 percentage expression determined by immunohistochemistry (IHC).

DETAILED DESCRIPTION:
A non-blinded, single centre, single interventional arm Phase II diagnostic imaging study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Patients with histopathology confirmed untreated metastatic NSCLC scheduled for systemic anti-cancer therapy
* ECOG status ≤ 1
* Willingness and ability to comply with scheduled study visits and tests

Exclusion Criteria:

* Pregnant or breast-feeding women
* Concomitant uncontrolled medical conditions as per Investigator assessment
* > 3 months between IHC PD-L1 and study recruitment
* Significant abnormality of haematology (one or more of: Hb ≤ 90g/L, absolute neutrophil count (ANC) ≤1.5 x109/L, platelet count ≤75 x109/L)
* Significant abnormality of renal function (defined as Cockcroft-Gault calculated creatinine clearance ≤30 mL/min)
* Significant abnormality of liver function (one or more of: AST or ALT ≥2.5x ULN or ≥ 5x ULN if patient has liver metastases; total bilirubin ≥1.5xULN. In the case of patients with Gilbert's syndrome then direct bilirubin must be confirmed as ≤ ULN)
* Significant cardiovascular disease, including New York Heart Association (NYHA) heart failure ≥Class III, myocardial infarction within 3 months of enrolment, unstable arrhythmia or unstable angina
* History of uncontrolled allergic reactions and/or have hypersensitivity to anti-PD-L1 monoclonal antibodies, kanamycin A or aminoglycoside therapies, or other excipients that may induce hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
PD-L1 Expression Assessment using [99mTc]-NM-01 SPECT/CT | Day 0
  To measure PD-L1 expression in NSCLC (primary tumour and metastatic lesions) as assessed using [99mTc]-NM-01 SPECT/CT and compare to PD-L1 expression determined by IHC.

SECONDARY OUTCOMES:
Safety of [99mTc]-NM-01 SPECT/CT assessed through incidence of Adverse Drug Reactions | Up to 12 days post-injection
  To assess the safety of [99mTc]-NM-01 SPECT/CT scan by observing for Adverse Drug Reactions (ADRs) occurring during the trial.
PD-L1 expression heterogeneity as assessed by [99mTc]-NM-01 SPECT/CT tumour to blood-pool ratios in each lesion | Day 0
  To measure intra-tumoural heterogeneity in the primary tumour, as well as in individual metastases and inter-tumoural heterogeneity between different disease sites (including different metastatic sites and between primary tumour and its metastases).

OTHER OUTCOMES:
Exploratory Objectives | Up to 16 weeks post-injection
  To correlate the SPECT/CT PD-L1 assessment with other diagnostic parameters such as blood tumour mutation burden test and to detect the presence of anti-drug antibodies to [99mTc]-NM-01.

CONTACTS AND LOCATIONS:
Overall Officials: Gary JR Cook, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust | King's College London, London, UK
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong NC, Cai Y, Meszaros LK, Biersack HJ, Cook GJ, Ting HH, Mottaghy FM. Preclinical development and characterisation of 99mTc-NM-01 for SPECT/CT imaging of human PD-L1. Am J Nucl Med Mol Imaging. 2021 Jun 15;11(3):154-166. eCollection 2021. PMID 34234994
- [Background] Xing Y, Chand G, Liu C, Cook GJR, O'Doherty J, Zhao L, Wong NCL, Meszaros LK, Ting HH, Zhao J. Early Phase I Study of a 99mTc-Labeled Anti-Programmed Death Ligand-1 (PD-L1) Single-Domain Antibody in SPECT/CT Assessment of PD-L1 Expression in Non-Small Cell Lung Cancer. J Nucl Med. 2019 Sep;60(9):1213-1220. doi: 10.2967/jnumed.118.224170. Epub 2019 Feb 22. PMID 30796165
- [Background] Hughes DJ, Chand G, Goh V, Cook GJR. Inter- and intraobserver agreement of the quantitative assessment of [99mTc]-labelled anti-programmed death-ligand 1 (PD-L1) SPECT/CT in non-small cell lung cancer. EJNMMI Res. 2020 Dec 1;10(1):145. doi: 10.1186/s13550-020-00734-x. PMID 33259032 (Retraction: PMID 34637006 EJNMMI Res. 2021 Oct 12;11(1):102)
- [Derived] Hughes DJ, Chand G, Johnson J, Bailey D, Adamson K, Goh V, Cook GJR. Inter-rater and intra-rater agreement of [99mTc]-labelled NM-01, a single-domain programmed death-ligand 1 (PD-L1) antibody, using quantitative SPECT/CT in non-small cell lung cancer. EJNMMI Res. 2023 May 31;13(1):51. doi: 10.1186/s13550-023-01002-4. PMID 37256434